CLINICAL TRIAL: NCT06947109
Title: A Phase I Clinical Study on Dose Escalation Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a Single Subcutaneous Dose of AK139 in Healthy Subjects.
Brief Title: A Clinical Study of AK139 in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK139-101
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK139 regimen (Active Comparator)
  Interventions: Drug: AK111
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Monitor for a minimum of 24 hours to assess whether the safety and tolerability are acceptable according to the investigator.
  Arms: Placebo
Drug: AK111 — The study will use dose escalation scheme. Before proceeding to randomize the next group of subjects, the safety data from all subjects in the previous dose group must be reviewed and confirmed.
  Arms: AK139 regimen

SUMMARY:
This is a phase I clinical study on dose escalation evaluating the safety, tolerability, PK and PD of a single dose of AK139 administered subcutaneously in healthy subjects.

DETAILED DESCRIPTION:
This is a phase I, dose escalation clinical study aimed to evaluate the safety, tolerability, PK and PD of AK139 in healthy subjects. This study will be conducted in a dose escalation design, sequentially increasing the dosage of the drug from low to high to complete a single subcutaneous dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily agree to participate and sign an informed consent form (ICF) before any study procedures begin.
* Male and female healthy subjects aged 18 to 55 at the time of signing the ICF.
* Male weight ≥ 50.0kg, female weight ≥ 45.0kg; Body Mass Index (BMI)=Weight (kg)/Height² (m²), within the range of 19.0~26.0 kg/m².
* Female subjects with fertility tested negative for pregnancy during the screening period.
* The subjects are able to communicate well with the investigator and understand and comply with the requirements of this study.

Exclusion Criteria:

* Allergies to AK139 components and any monoclonal antibodies.
* Positive results of confirmatory serology test for hepatitis B, hepatitis C,HIV or syphilis at screening.
* have participated in any drug clinical study within 3 months prior to randomization, or are still within 5 half-lives after the last administration of other investigational drugs (whichever is longer)
* Previously or currently suffering from any diseases of the circulatory, endocrine, neurological, digestive, respiratory, urogenital, blood, immune, psychiatric, or metabolic systems that may interfere with the test results.
* History of parasitic infection.
* Drug abusers or individuals with positive urine drug results during screening.
* Have donated blood or experienced significant blood loss, received blood transfusions, or used blood products 3 months before screening.
* Investigator assessed that it is not suitable to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-05-06 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) | Baseline to week 12
  The incidence of AEs . An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.

SECONDARY OUTCOMES:
Peak concentration (Cmax) | Week 0 to week 12
  Measure and assess the Cmax of AK139.
Time to peak (Tmax) | Week 0 to week 12
  Measure and assess the Tmax of AK139
Area under the curve (AUC) | Week 0 to week 12
  Measure and assess the AUC of AK139
Half-life (t1/2) | Week 0 to week 12
  Measure and assess the t1/2 of AK139.
Anti-drug antibody (ADA) | Week 0/2/4/8/12
  Measure and assess the ADA of AK139.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Xiaoshan Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No